CLINICAL TRIAL: NCT04954274
Title: Improvement of Live Babies Rates After ICSI, Using cpFT: Multicenter Prospective Randomized Clinical Trial
Brief Title: Improvement of Live Babies Rates After ICSI, Using cpFT
Acronym: FERTICSI
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P170706J
Record Dates: First submitted 2021-04-29; First posted 2021-07-08 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Infertility; Oocyte; Pregnancy
Keywords: Infertility; Femal infertility; Assisted Reproduction Technology outcome
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: there will be two groups: one treated by supplementation of the culture medium with 1 Micromolar of the molecule, the other being the control group.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fertiline group (Experimental): Treated by supplementation of the culture medium with the molecule.
  Interventions: Drug: Cyclic peptide Fertiline
- Control group (No Intervention): No supplementation

INTERVENTIONS:
Drug: Cyclic peptide Fertiline — Upon retrieval, the oocyte will be decoronized and incubated prior to ICSI procedure into CSCC-M medium supplemented with the molecule.
  After ICSI, the zygote will be incubated in CSCM-C medium supplemented with the peptide.
  Other Names: cFEE
  Arms: Fertiline group

SUMMARY:
Demonstrate the improvement of the live births rate after ICSI by supplementing the pre-ICSI incubation medium of oocytes and that of preimplantation embryos with cpFT at the 1st embryo transfer for women under 37 years old.

DETAILED DESCRIPTION:
Supplementation of the incubation medium with cFEE should improve the implantation rate and ART outcome.

As in France ICSI is widely used to achieve good fertilization rates, we decided to use ICSI to fertilize the egg, and the peptide:

1. to improve chromosome segregation during meiosis, and
2. to improve in vitro embryogenesis after ICSI. Hence the protocol includes an oocyte preincubation step prior to ICSI and a co incubation of the embryo with the molecule during blastocyst formation.

Hence our protocol includes:

1. - a preincubation of the decoronized oocytes with the peptide prior to ICSI, and
2. - a coincubation of the developing embryo with the molecule.

The principal criteria will be the live baby rate after the first embryo transfer (using the best embryo). As the oocyte loses its strength as the women is getting older, the main criteria will be evaluated for women under 37 years old.

Randomization: every couple will be randomly assigned to the Control or the Treated group.

Treated group: After egg retrieval, the oocyte will be decoronized and incubated prior to ICSI procedure into CSCM-C (Irvine) medium supplemented with the molecule.

Control group: similar protocol of incubation but without the molecule. After ICSI the zygote will be incubated until the blastocyste stage in CSCM-C medium (Irvine).

Embryo transfer will be limited to only one blastocyst, fresh or delayed after cryopreservation.

ELIGIBILITY:
Inclusion Criteria:

* Couples eligible for a attempt at Assisted Reproduction (AMP).
* Couples asking for Assisted Reproductive Technology, and requiring an ICS procedure.
* Women aged 18 to 36 inclusive.
* Men aged 18 to 58 inclusive
* Use of CSCM-C culture medium from Biocare / Irvine, exclusively.
* People affiliated to a Social Security scheme

Exclusion Criteria:

* Lack of consent
* Early menopause.
* Couples under IVF or Intra Uterine Insemination treatment.
* People unable to follow protocol visits in France.
* Couple with a contraindication to treatment with ART.
* Women with a contraindication to treatment with ART or an associated pathology such as: hypertension, risk of eclampsia, family genetic problems, diabetes, uterine partitions, synechiae adhesions, adenomyosis or any other contraindication judged as such by the investigator.
* ART with donation of gametes or embryos.
* Participant under guardianship or guardianship

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 366 (Estimated)
Dates: Start 2021-07-29 (Actual); Primary Completion 2026-07-29 (Estimated); Study Completion 2027-07-29 (Estimated)

PRIMARY OUTCOMES:
Live birth rate after the first embryo transfer | 54 months after the first randomization
  Demonstration of the improvement in the rate of live births after ICSI by supplementing the pre-ICSI incubation medium of oocytes and that of preimplantation embryos with cpFT (1µM) during the 1st embryo transfer in women under 37 years of age.

SECONDARY OUTCOMES:
Level of Metaphase II oocytes | During the randomization period, which is 42 months.
Quality of the embryonic culture | 42 months after the first randomization
  The measure evaluates the rate and number of fertilized eggs over the total number of metaphase 2 oocytes.
Evaluation of the kinetics of embryonic development when possible. | 42 months after the first randomization
  The embryos will be kept in an incubator with an embryoscope so that their cleavage sequences will be registered "when possible". The criteria will analyze the cleavage sequence of all embryos during preimplantation embryogenesis.
Embryonic quality at the blastocyst stage | Day 5-6 after ICSI
  All the embryos that will reach the blastocyst stage will be evaluated according to the Gardner criteria.
Quality of the embryos after vitrification | Day 5-6 after ICSI
  The percentage of Good and Top embryos after thawing will be compared to the grading for the same embryo before cryopreservation according to Gardner criteria
Implantation rate with positive Beta hCG after transfer | 54 months after the first randomization
  This criterion will be evaluated only for the first embryo transfer of each enrolled couple.
Clinical pregnancy rates with cardiac activity | until 54 months after the first randomization
  This criterion will be evaluated only for the first embryo transfer of each enrolled couple.
The rate of miscarriages per pregnancy | until 54 months after the first randomisation
  This criterion will be evaluated only for the first embryo transfer of each enrolled couple.
rate of abnormality on morphological ultrasounds | 51 months after the first randomisation
  It reports the percentage of morphological ultrasounds showing an abnormality in the fetus morphology on the total number of morphological ultrasounds performed for all the pregnancies depending of the study.
  This creterion will be assessed for all transfers that occurred during the randomization period and for the following 3 months in the case of deferred transfers.
rate of neonatal abnormality | 54 months after the first randomisation
  It reports the percentage of neonatal baby examination showing an abnormality over the total number of neonatal baby examination performed for all the babies who will born during the study.
  This criterion will be assessed for all transfers that occurred during the randomization period and for the following 3 months in the case of deferred transfers.
children's development | 72 months after the beginning of the study
  It reports the percentage of one year old baby examinations showing an abnormality over the total number of one year old baby examinations performed for all the babies who will born during the study.
  This criterion will be assessed for all transfers that occurred during the randomization period and for the following 3 months in the case of deferred transfers.
Weight of the placenta; Study of DNA, RNA, Western-Blot, Methylation, histological study | 54 months after the first randomization
  This outcome concerns patientes who give birth in the maternity ward of the Cochin hospital

CONTACTS AND LOCATIONS:
Overall Officials: Jean Philippe Mr WOLF, MD-PhD, Principal Investigator — AP-HP, Hospital Cochin
Locations (1):
- Department Biology of Reproduction, Hospital Cochin AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barraud-Lange V, Naud-Barriant N, Ducot B, Chambris S, Bomsel M, Wolf JP, Ziyyat A. Cyclic QDE peptide increases fertilization rates and provides healthy pups in mouse. Fertil Steril. 2009 May;91(5 Suppl):2110-5. doi: 10.1016/j.fertnstert.2008.05.088. Epub 2008 Aug 9. PMID 18692807
- [Background] Ziyyat A, Naud-Barriant N, Barraud-Lange V, Chevalier F, Kulski O, Lemkecher T, Bomsel M, Wolf JP. Cyclic FEE peptide increases human gamete fusion and potentiates its RGD-induced inhibition. Hum Reprod. 2005 Dec;20(12):3452-8. doi: 10.1093/humrep/dei241. Epub 2005 Aug 11. PMID 16096325